CLINICAL TRIAL: NCT07112716
Title: Superior Vena Cava Isolation With Radiofrequency Ablation in Patients With Recurrent Paroxysmal Atrial Fibrillation and Durably Isolated Pulmonary Veins: A Multicenter Study
Brief Title: SVC-isolation in Redo-AF Ablation With Isolated PV
Acronym: SVC-RESCUE-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, MD, PhD, Centro Medico Teknon
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVC-RESCUE-AF; SVC-RESCUE-AF (Other: Teknon Medical Centre)
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Paroxysmal AF
Keywords: Atrial fibrillation; Paroxysmal; Recurrence; Superior Vena Cava Isolation
MeSH Terms: conditions — Atrial Fibrillation; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SVC isolation group (Active Comparator): Empirical superior vena cava isolation
  Interventions: Procedure: Empirical superior vena cava isolation
- Control arm (Sham Comparator): No empirical superior vena cava isolation
  Interventions: Procedure: Ablation without empirical superior vena cava isolation

INTERVENTIONS:
Procedure: Empirical superior vena cava isolation — Empirical superior vena cava isolation with radiofrequency ablation
  Arms: SVC isolation group
Procedure: Ablation without empirical superior vena cava isolation — No ablation or ablation of other arrhythmic foci wuthout empirical superior vena cava isolation
  Arms: Control arm

SUMMARY:
Atrial fibrillation is the most common arrhythmia in the population and is often caused by arrhythmogenic foci located in the pulmonary veins. For this reason, the first attempt in atrial fibrillation catheter ablation procedures is to isolate these structures (the procedure is called indeed "pulmonary vein isolation"), which results in abolishment of arrhythmia recurrence in up to 85% of patients at short and mid-term follow-up. However, a subset of patients experience an atrial tachyarrhytmia recurrence and a second catheter ablation procedure has to be performed. If pulmary vein isolation is proven to be durable, other arrhythmogenic foci could be implicated in arrhythmia recurrence. Among extra-pulmonary vein foci, superior vena cava has been described as the most frequently involved in atrial fibrillation initiation. Therefore, its ablation could result in improved freedom from atrial fibrillation episodes during follow-up. In the present study, we sought to evaluate the safety and effectiveness of empirical superior vena cava isolation in terms of arrhythmia-free survival in patients with paroxysmal atrial fibrillation recurrence despite durable pulmonary vein isolation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most frequent arrhythmia in the general population (1), with an expected doubling in prevalence within 2060 (2). Since the late 1990s (3), pulmonary vein isolation (PVI) has become a cornerstone in drug refractory AF treatment, and more recently has emerged a first line therapy in paroxysmal AF patients (4) due to its proven superiority to antiarrhythmic drugs in achieving arrhythmia-free survival (5).

PVI is a safe and effective procedure in the vast majority of patients with paroxysmal AF, with high AF-free survival at mid- and long-term follow-up. In case of AF recurrence, repeat ablation of pulmonary vein reconnections demonstrated superior outcomes compared to the use of anti-arrhythmic drugs in both paroxysmal and persistent AF (6). Nevertheless, a subset of patients with AF recurrence results to be "PVI non-responder", with arrhythmia recurrence despite durable ablation results (7). How to manage these patients is still a matter of debate, with different additional lesion sets proposed so far (8).

Non-PVI triggers have been implicated in AF initiation, with superior vena cava (SVC) being the most common of them (9,10). Empirical SVC isolation has been attempted in some observational as well as randomized study (11-14), but definitive conclusion could not be drawn due to lack of statistical power as well as variable eligibility criteria (first vs repeat procedure, paroxysmal vs persistent AF) and ablation sets (15).

In the present study, we sought to evaluate the safety and effectiveness of empirical SVC isolation in terms of arrhythmia-free survival in patients with paroxysmal AF recurrence despite durable PVI.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Confirmed diagnosis of recurrent paroxysmal AF
3. Previous transcatheter PVI-only procedure for AF.
4. Evidence of persistently isolated pulmonary veins at repeat procedure.
5. Signed informed consent.

Exclusion Criteria:

* Age < 18 years.
* Pregnancy.
* Concomitant investigation treatments.
* Medical, geographical and social factors that make study participation impractical, and inability to give written informed consent. Patient's refusal to participate in the study.
* Lesions other than PVI performed during first procedure
* Persistent AF at recurrence.
* Evidence of pulmonary vein reconnection at repeat procedure.
* Any additional lesion performed beyond SVC isolation during repeat procedure (in the empirical SVC isolation group only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Arrhythmia-free survival | 12 months follow-up
  Occurence of any sustained atrial arrhythmia (AF, atrial flutter or any atrial tachycardia) lasting ≥ 30 s, after a 2-month blanking period

SECONDARY OUTCOMES:
Procedure-related complications | 12 months follow-up
  Any procedure complication

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Berruezo, MD, PhD, Principal Investigator — Teknon Medical Centre
Locations (1):
- Heart Institute, Teknon Medical Centre, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided